CLINICAL TRIAL: NCT00391248
Title: A Phase II Trial of Erlotinib and Concurrent Palliative Thoracic Radiation Therapy for Patients With Non-small Cell Carcinoma of the Lung. (PEARL Trial)
Brief Title: Phase II Trial of Erlotinib and Concurrent Palliative Thoracic Radiation Therapy for Non-small Cell Lung Cancer (PEARL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTA-Control-105472
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2011-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; palliative radiation; tarceva; palliative thoracic radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Erlotinib — 150 mg in a single daily dose, starting Day 1 through Day 22
  Other Names: Tarceva

SUMMARY:
To improve the clinical outcomes of patients with non-small cell lung cancer treated with radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (squamous cell, adenocarcinoma, poorly differentiated non-small cell carcinoma, or some combination of these); and
* Symptomatic patients (defined at discretion of investigator) for whom palliative thoracic radiation is planned (3000cGy/10 fractions); and
* At least 18 years of age.

Exclusion Criteria:

* Previous erlotinib therapy; or
* Planned concurrent chemotherapy; or
* Expected survival of less than 3 months; or
* ECOG Performance Status of 3 or 4; or
* Multiple CNS metastasis or a single CNS lesion that has not demonstrated radiologic stability (screening CT/MRI or head not required); or
* Granulocyte count <1,500/mm3, platelet count <100,000/mm3, or haemoglobin <9.0g/dl; or
* SGOT (AST) or SGPT (ALT) > 2.5 times (x) upper limit of normal (ULN) in the absence of known liver metastases or > 5 x ULN in case of known liver metastases; or
* Alkaline phosphatase (ALP) > 2.5 x ULN; or
* Serum bilirubin > 1.5 ULN; or
* Serum creatinine > 1.5 ULN or creatinine clearance < 60 ml/min; or
* Serum calcium beyond ULN; or
* Patients requiring systemic anti-fungal therapy, clarithromycin, phenytoin, or oral anticoagulation therapy (see Appendix VI for complete list of medications); or
* A history of interstitial lung disease; or
* Known sensitivity to erlotinib; or
* Pregnancy, lactation, or parturition within the previous 30 days; or
* Unwillingness or inability to complete the required assessments of the trial; or
* Mental incompetence, including psychiatric or addictive disorders which would preclude meaningful informed consent; or
* History of recurrent conjunctivitis or keratitis or other inflammatory changes of the surface of the eye.
* Geographically inaccessible for treatment or follow-up evaluations; or
* Involved in an ongoing therapeutic trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The mean improvement of "lung cancer symptoms" as measured by the Lung Cancer Symptom Scale at four weeks following completion of radiation therapy | 4 weeks post radiotherapy

SECONDARY OUTCOMES:
The improvement in global quality of life and total scores of the LCSS at four weeks following treatment, radiological response, and the incidence and severity of adverse events as per the CTCAE version 3 | 4 weeks post radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jim Wright, MD, Principal Investigator — Juravinski Cancer Centre
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario